CLINICAL TRIAL: NCT07090330
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of ORKA-001 in Participants With Moderate-to-Severe Plaque Psoriasis
Brief Title: ORKA-001 Versus Placebo in Patients With Moderate-to-Severe Plaque Psoriasis
Acronym: EVERLAST-A
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oruka Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORKA-001-112
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Plaque Psoriasis
Keywords: Phase 2; ORKA-001; Plaque psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- (Induction Period) ORKA-001 (Experimental): Participants will receive ORKA-001 per protocol Induction regimen.
  Interventions: Drug: ORKA-001 Induction Dose
- (Induction Period) Placebo (Placebo Comparator): Participants will receive Placebo per protocol Induction regimen.
  Interventions: Other: Placebo
- (Maintenance Period - Arm 1) ORKA-001 (Experimental): Participants will receive ORKA-001 per protocol Maintenance regimen, based on protocol defined response.
  Interventions: Drug: ORKA-001 Maintenance Dose
- (Maintenance Period - Arm 2) ORKA-001 (Experimental): Participants will receive ORKA-001 per protocol Maintenance regimen, based on protocol defined response.
  Interventions: Drug: ORKA-001 Maintenance Dose
- (Maintenance Period - Arm 3) Placebo (Placebo Comparator): Participants will receive Placebo per protocol Maintenance regimen, based on protocol defined response.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ORKA-001 Induction Dose — ORKA-001 Induction Dose, administered by subcutaneous (SC) injection
  Arms: (Induction Period) ORKA-001
Other: Placebo — Placebo administered by subcutaneous (SC) injection
  Arms: (Induction Period) Placebo; (Maintenance Period - Arm 3) Placebo
Drug: ORKA-001 Maintenance Dose — ORKA-001 Maintenance Dose, administered by subcutaneous (SC) injection
  Arms: (Maintenance Period - Arm 1) ORKA-001; (Maintenance Period - Arm 2) ORKA-001

SUMMARY:
This is a multicenter, randomized, double-blinded, placebo-controlled, proof-of-concept study to evaluate the efficacy, safety, tolerability, and pharmacokinetics of ORKA-001 in adult participants with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a proof-of-concept study evaluating ORKA-001 in patients with moderate-to-severe psoriasis with study drug administration divided into an Induction period followed by a Maintenance period. Following completion of the Maintenance period at Week 52, participants will have the option to enter into the open-label extension (OLE) study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥ 18 years of age
2. Have a diagnosis of plaque psoriasis for > 6 months
3. Have moderate-to-severe chronic plaque psoriasis defined as:

   1. BSA ≥ 10%, and
   2. PASI ≥ 12, and
   3. IGA score of ≥ 3 on a 5-point scale
4. Candidate for systemic therapy or phototherapy
5. Women of childbearing potential must have a negative pregnancy test

Exclusion Criteria:

1. Nonplaque forms of psoriasis (including guttate, erythrodermic, or pustular) or drug-induced psoriasis
2. Significant history or clinical manifestation of any metabolic, other dermatological, hepatic, renal, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, respiratory, endocrine, or psychiatric disorder, or any infectious disease
3. History of malignancy, except for non-melanoma skin cancer or cancer curatively treated ≥ 5 years, without evidence of recurrence
4. A known hypersensitivity to any components of the ORKA-001 drug product
5. Women who are breastfeeding or plan to breastfeed during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving 100% Reduction in PASI Score at Week 16 | Week 16
  The Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).

SECONDARY OUTCOMES:
Proportion of Participants Who Achieve an IGA = 0 (Clear) at Week 16 | Week 16
  The Investigator Global Assessment (IGA) documents the Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Proportion of Participants Achieving 90% Reduction in PASI Score at Week 16 | Week 16
  Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).
Proportion of Participants Who Achieve an IGA = 0 (Clear) or 1 (Almost Clear) at Week 16 | Week 16
  The Investigator Global Assessment (IGA) documents the Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Proportion of Participants Maintaining 100% Reduction in PASI Score at Week 52 | Week 52
  The Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).
Proportion of Participants Maintaining an IGA = 0 (Clear) at Week 52 | Week 52
  The Investigator Global Assessment (IGA) documents the Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Proportion of Participants Maintaining 90% Reduction in PASI Score at Week 52 | Week 52
  The Psoriasis Area and Severity Index Score (PASI) is an evaluation tool that combines the assessment of the severity and the area affected by psoriasis into a single score ranging from 0 (no disease) to 72 (maximum disease).
Proportion of Participants Maintaining an IGA = 0 (Clear) or 1 (Almost Clear) at Week 52 | Week 52
  The Investigator Global Assessment (IGA) documents the Investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as clear (0), almost clear (1), mild (2), moderate (3), or severe (4).
Incidence of Treatment-emergent Adverse Events | Day 1 through 52 Weeks
  Incidence of treatment adverse events and clinically significant changes from baseline in vital signs, clinical laboratory parameters and electrocardiograms

CONTACTS AND LOCATIONS:
Locations (24):
- United States (16):
  - Oruka Therapeutics Investigative Site, Fountain Valley, California
  - Oruka Therapeutics Investigative Site, Los Angeles, California
  - Oruka Therapeutics Investigative Site, San Diego, California
  - Oruka Therapeutics Investigative Site, Santa Ana, California
  - Oruka Therapeutics Investigative Site, Santa Monica, California
  - Oruka Therapeutics Investigative Site, Cromwell, Connecticut
  - Oruka Therapeutics Investigative Site, Coral Gables, Florida
  - Oruka Therapeutics Investigative Site, Rolling Meadows, Illinois
  - Oruka Therapeutics Investigative Site, Bowling Green, Kentucky
  - Oruka Therapeutics Investigative Site, Rockville, Maryland
  - Oruka Therapeutics Investigative Site, Boston, Massachusetts
  - Oruka Therapeutics Investigative Site, Detroit, Michigan
  - Oruka Therapeutics Investigative Site, New York, New York
  - Oruka Therapeutics Investigative Site, Portland, Oregon
  - Oruka Therapeutics Investigative Site, Norfolk, Virginia
  - Oruka Therapeutics Investigative Site, Milwaukee, Wisconsin
- Canada (8):
  - Oruka Therapeutics Investigative Site, Edmonton, Alberta
  - Oruka Therapeutics Investigative Site, Surrey, British Columbia
  - Oruka Therapeutics Investigative Site, Hamilton, Ontario
  - Oruka Therapeutics Investigative Site, London, Ontario
  - Oruka Therapeutics Investigative Site, Markham, Ontario
  - Oruka Therapeutics Investigative Site, Peterborough, Ontario
  - Oruka Therapeutics Investigative Site, Toronto, Ontario
  - Oruka Therapeutics Investigative Site, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: Undecided